CLINICAL TRIAL: NCT03418415
Title: Renal Denervation in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Clinical Professor, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018RDN-T2DM
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes Mellitus; Renal Denervation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal denervation (Experimental): Procedure: Renal denervation
  Interventions: Device: Renal denervation

INTERVENTIONS:
Device: Renal denervation — multi-electrode catheter-based renal denervation

SUMMARY:
Sympathetic overactivity induces insulin resistance and type 2 diabetes mellitus (T2DM), so we assume that renal denervation (RDN) might improve glucose metabolism and insulin sensitivity. The purpose of this study is to evaluate the effects of multi-electrode catheter-based RDN on glucose metabolism and insulin sensitivity in patients with T2DM.

DETAILED DESCRIPTION:
Sympathetic overactivity induces insulin resistance and type 2 diabetes mellitus (T2DM), so it is assumed that renal denervation (RDN) might improve glucose metabolism and insulin sensitivity. Some clinical studies have shown that glucose metabolism is improved in patients with resistant hypertension both 1 and 3 months after RDN, and fasting glucose, insulin and C-peptide decreased significantly as did insulin resistance assessed by HOMA-IR. But in some clinical studies, RDN did not lead to a significant improvement of insulin sensitivity ≤12 months after treatment, and no effect in systemic sympathetic activity was observed after RDN. Therefore, the efficacy of RDN on glucose metabolism is still in controversy. The investigators wish to investigate the effect of multi-electrode catheter-based RDN on glucose metabolism and insulin sensitivity in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years and ≤ 70 years old
* Able and willing to provide informed consent
* Patients with established type II diabetes mellitus (HbA1C>7.5%, diet or oral hypoglycaemic agents)
* Clinical stable as demonstrated by no change in background anti-diabetic medication in the last 30 days.
* Anticipated that patients are able to maintain a stable dose of medication for the duration of the study

Exclusion Criteria:

* Renal arterial anatomy ineligible for RDN: main renal arteries <4 mm in diameter or <20 mm in treatable length; multiple renal arteries where main renal artery is estimated to supply <75% of the kidney
* History of prior renal artery intervention including balloon angioplasty, stenting or previous renal denervation
* Type 1 diabetes mellitus
* Pregnant, nursing or planning to be pregnant
* Orthostatic hypotension
* eGFR <30 ml/min (MDRD formula)
* Patients that have allergy to contrast agent
* Myocardial infarction, unstable angina pectoris, coronary bypass or percutaneous angioplasty within 3 months before inclusion
* Cerebrovascular accidents and alimentary tract hemorrhage within 3 months before inclusion
* Any medical condition which, in the investigators opinion, may adversely affect the participants safety in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Changes in glucose metabolism from baseline to 6 months | 6 months
  To investigate the influence of RDN on glucose metabolism. Hereby evaluating Oral Glucose Tolerance Test (OGTT) and glycosylated hemoglobin (HbA1c) before and after RDN.

SECONDARY OUTCOMES:
Changes in glucose metabolism up to 2 years | 3, 12 and 24 months
  To investigate the influence of RDN on glucose metabolism. Hereby evaluating Oral Glucose Tolerance Test (OGTT) and glycosylated hemoglobin (HbA1c) before and after RDN.
Changes in insulin and C-peptide up to 2 years | 3, 6, 12 and 24 months
  To investigate the influence of RDN on insulin and C-peptide.
Changes in catecholamine up to 2 years | 3, 6, 12 and 24 months
  To investigate the influence of RDN on catecholamine.
Changes in glucagon up to 2 years | 3, 6, 12 and 24 months
  To investigate the influence of RDN on glucagon.
Changes in blood pressure up to 2 years | 3, 6, 12 and 24 months
  To investigate the influence of RDN on blood pressure.
Changes in triglyceride and high density lipoprotein (HDL) up to 2 years | 3, 6, 12 and 24 months
  To investigate the influence of RDN on triglyceride and HDL.
Changes in renal function up to 2 years | 3, 6, 12 and 24 months
  To investigate the influence of RDN on creatinine and blood urea nitrogen (BUN).

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No